## Title: A Novel Approach for Brain Stimulation in Severe Stroke NCT03868410

10/23/24

**Statistical Analysis Summary for Results** 

## Statistical Analysis Plan\_Results

Statistical analysis was performed in R 4.3.1. Shapiro-Wilks tests were used to evaluate normality of data. For each motor outcome measure, we used repeated-measures ANOVA or Friedman's test to evaluate whether the outcome changed across time, separately for each group. When the omnibus test was statistically significant, post hoc pairwise comparisons were carried out using paired t-tests or Wilcoxon signed-rank tests, and multiple comparisons were corrected using the Holm-Bonferroni method. To understand whether treatment effects differed between groups, we used independent t-tests or Wilcoxon rank sum tests to compare change scores between groups. Because we did not find any change between post-test and follow-up timepoints in either group, we focused between-group comparisons on change from pre-test to post-test and change from pre-test to follow-up. The Holm-Bonferroni method was used to correct for multiple comparisons.

For TMS outcomes, we used paired t-tests or Wilcoxon signed rank tests to evaluate whether each outcome changed across time, separately for each group. To understand whether treatment effects differed between groups, we compared change scores between groups with Wilcoxon rank sum tests. We also explored whether change in motor function (motor outcomes) were associated with change in TMS.